CLINICAL TRIAL: NCT04870762
Title: A Randomized Study of Head and Neck Radiotherapy With or Without Customized 3D Printed Oral Stents
Brief Title: Customized 3D Printed Oral Stents During Head and Neck Radiotherapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-1153; NCI-2021-03221 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-1153 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-04-23; First posted 2021-05-03 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Head and Neck Carcinoma; Malignant Parotid Gland Neoplasm; Maxillary Sinus Carcinoma; Nasal Cavity Carcinoma; Oral Cavity Carcinoma; Tongue Carcinoma; Tonsillar Carcinoma
MeSH Terms: conditions — Parotid Neoplasms; Maxillary Sinus Neoplasms; Mouth Neoplasms; Tongue Neoplasms; Tonsillar Neoplasms | interventions — Practice Guidelines as Topic; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Arm I (3D printed oral stent) (Experimental): Patients wear 3D printed oral stent during standard of care radiotherapy.
  Interventions: Other: Best Practice; Other: Medical Device Usage and Evaluation
- Arm II (standard of care) (Active Comparator): Patients receive standard of care during treatment.
  Interventions: Other: Best Practice; Other: Medical Device Usage and Evaluation

INTERVENTIONS:
Other: Best Practice — Receive standard of care
  Other Names: standard of care; standard therapy
Other: Medical Device Usage and Evaluation — Wear 3D printed oral stent

SUMMARY:
This clinical trial studies the effect of customized 3 dimensional (3D) printed oral tents on patients with head and neck cancer who are receiving radiotherapy. Oral stents are made from the impression of patients' mouth and cover patients' teeth and gums during radiation therapy. A customized, 3D-printed oral stent may help to reduce mouth blisters and/or sores that may develop in patients while receiving head and neck radiation therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the acute mucositis rates in non-target mucosa of patients who receive head and neck radiation with or without a customized 3D printed oral stent.

SECONDARY OBJECTIVES:

I. To record patient reported outcomes during radiotherapy. II. To evaluate patient narcotic use during radiotherapy. III. To evaluate the imaging and dosimetric differences in head and neck radiotherapy with and without a customized 3D printed oral stent.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients wear 3D printed oral stent during standard of care radiotherapy.

ARM II: Patients receive standard of care during treatment.

ELIGIBILITY:
Inclusion Criteria:

* Participant is dispositioned to receive 5-7 weeks of definitive or adjuvant radiotherapy for treatment of a diagnosed head and neck malignancy
* Age 18 or older
* ECOG PS 0-2
* The participant will receive either (a) radiation alone or (b) radiation with concurrent chemotherapy of any kind(s)
* Signed study-specific consent form

Exclusion Criteria:

* Prior head and neck radiotherapy
* Participants is unable to fit a tongue-lateralizing or tongue-depressing stent
* Severe trismus with an incisal opening of <10 mm
* Inability to comply with the study procedures
* Participants younger than 18 years of age
* Participants must not be pregnant
* Cognitively impaired subjects

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Estimated)
Dates: Start 2021-05-26 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Mucositis toxicity rates | Through study completion, an average of 1 year
  Rate of non-target mucose will be estimated along with the corresponding 95% confidence interval. Cochran-Mantel-Haenszel (CHM) test will be applied to compare mucositis rates between the two treatment arms. Logistic regression will be used to compare occurrence of mucositis between two arms, adjusting for the effects of stratification factors as well as other covariates. T test or Wilcoxon rank sum test will be used to compare three Olerud-Molander Ankle Score between two arms: a mean mucositis score, an extent of mucositis score, and a worst site score.

SECONDARY OUTCOMES:
Patient reported outcomes | Through study completion, an average of 1 year
  Will be assessed using the MD Anderson Symptom Inventory Head and Neck questionnaire. T test or Wilcoxon rank sum test will be used to compare scores of each item per time point or sums of scores across all items at each time point or sums across three time point per item between the two arms. Multivariate analyses such as linear regression model adjusting for the effects of covariates might be performed to compare patients reported outcomes. Appropriate data transformation will be performed if necessary for assumption of normality.
Patients narcotics diaries | Through study completion, an average of 1 year
  Will record the worst, the least, the average pain score and pain score at present for each day. Will calculate the average of these 4 scores as a composite daily pain score.
Imaging difference | Through study completion, an average of 1 year
  The set up error during radiation will be measured in each treatment arm.
Dosimetric difference | Through study completion, an average of 1 year
  The radiation dose to healthy tissue will be measured in each treatment arm.
Composite pain scores | Through study completion, an average of 1 year
  An area under curve of pain scores over two weeks (AUC2wks) will be calculated for each patient, and the t test or Wilcoxon rank sum test will be used to compare the AUC2wks of pain scores between the two arms, and between patients with and without occurrence of mucositis in their non-target mucosa. Will also fit linear mixed models including patients as random effects to compare the composite pain scores over two weeks between treatment arms. The linear mixed models will also be fitted to evaluate the association of composite pain scores with occurrence of their non-target mucosa.
Number of narcotic pills used | Through study completion, an average of 1 year
  An AUC2wks will be calculated for each patient, and the t test or Wilcoxon rank sum test will be used to compare the AUC2wks of pain scores between the two arms, and between patients with and without occurrence of mucositis in their non-target mucosa. Will also fit linear mixed models including patients as random effects to compare the composite pain scores over two weeks between treatment arms.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Lee, Principal Investigator — M.D. Anderson Cancer Center
Locations (7):
- United States (7):
  - Banner Health/Banner Research, Phoenix, Arizona
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - Community MD Anderson Cancer Center East, Indianapolis, Indiana
  - Community MD Anderson Cancer Center South, Indianapolis, Indiana
  - Community MD Anderson Cancer Center North, Indianapolis, Indiana
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - M D Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org